CLINICAL TRIAL: NCT01902823
Title: Pilot Test of the Effect of Cancer Nurse Navigators on Patient Outcomes
Brief Title: Effect of Cancer Nurse Navigators on Patient Outcomes
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Clinicians were not offering the study to eligible potential subjects.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-86E; OS11336 (Other: UW Carbone Cancer Center); A545000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison)
Record Dates: First submitted 2011-11-29; First posted 2013-07-18 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-11

CONDITIONS: Lung Cancer; Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: Nurse Navigator; Satisfaction with Care; Quality of Life; Symptom Distress
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Nurse Navigator Services (No Intervention)
- Services from a Nurse Navigator (Experimental)
  Interventions: Behavioral: Services from a Nurse Navigator

INTERVENTIONS:
Behavioral: Services from a Nurse Navigator — Services from a Nurse Navigator
  Arms: Services from a Nurse Navigator

SUMMARY:
There is widespread anecdotal evidence that Cancer Nurse Navigators (CNNs) are highly valued by cancer patients, but no studies have evaluated the effects of CNNs on important patient-reported outcomes or indicators of quality of care. This study has two aims:

1. To assess the feasibility of studying the impact of Aurora CNN Program.
2. To pilot test the effects of CNN services on patient-reported outcomes and indicators of quality of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years of age or older)
2. Treated at Aurora St. Luke's or West Allis Medical Center
3. New or recurrent dx of lung, prostate, colorectal or breast cancer -

Exclusion Criteria:

1. Previously received CNN services at an Aurora treatment facility
2. Unable to read/write in English
3. Living in a nursing home/long term care facility
4. Not capable of completing study questionnaires -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Care | Change from baseline, to 3 months to 6 months

SECONDARY OUTCOMES:
ED/Urgent care visits | Baseline, 3 months, 6 months
Quality of Life | Baseline, 3 months, 6 months
  The Functional Assessment Cancer Therapy - General (FACT-G) assesses quality of life.
Distressed mood | Baseline, 3 months, 6 months
  The National Comprehensive Cancer Network Distress Thermometer assesses level of distress.
Symptom Distress | Baseline, 3 months, 6 months
  The Memorial Symptom Assessment Scale measures 32 common physical and psychological cancer-related symptoms.
The Inventory of Recent Life Experiences for Cancer Patients | Baseline, 3 months, 6 months
  This instrument measures 30 cancer-related irritants (hassles) commonly experienced by persons with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Kwekkeboom, PhD, RN, Principal Investigator — University of Wisconsin, Madison; Sandra E Ward, PhD, RN, Principal Investigator — Uniuversity of Wisconsin Madison
Locations (2):
- United States (2):
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin
  - Aurora West Allis, West Allis, Wisconsin